CLINICAL TRIAL: NCT02954042
Title: Pelvital Stress Urinary Incontinence Training Device: P-SUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pelvital USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: URO-2016-25004
Record Dates: First submitted 2016-10-28; First posted 2016-11-03 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Incontinence
Keywords: Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Pelvital probe (Experimental): Probe to use for incontinence-Pevital is company name of product
  Interventions: Device: Pelvital probe
- Placebo Probe (Placebo Comparator): Placebo probe
  Interventions: Device: Placebo Probe

INTERVENTIONS:
Device: Pelvital probe — Pelvital probe
  Arms: Pelvital probe
Device: Placebo Probe — Placebo Probe
  Arms: Placebo Probe

SUMMARY:
The purpose of this investigation is to compare the clinical benefits of using the Pelvital product, in comparison to a sham procedure as a noninvasive treatment for female incontinence

DETAILED DESCRIPTION:
120 subjects with SUI will be recruited into a randomized, double-blind, sham-controlled crossover trial. Subjects will be allocated in a 1:1 ratio (60 per arm) to either the control arm (PFMT) or the treatment arm (PFMT in conjunction with the Pelvital therapy). Subjects will conduct their respective therapy five minutes a day over the course of six weeks. At weeks two, four and six, the subjects will conduct bi-weekly check-ups. After six weeks, all patients in the control arm will have the option to cross over into the treatment arm if no improvement in symptoms has been shown.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender,
2. Ages 18-75,
3. Clinical diagnosis of stress urinary incontinence,
4. Ability to contract the pelvic floor muscles,
5. Able to document incontinence and voiding in a diary,
6. Provision of written informed consent form,
7. Minimum of 10 grams increase at initial 24-hour pad weight test

Exclusion Criteria:

1. Diagnosed mixed or urge urinary incontinence,
2. Impaired cognitive function or neurologic conditions
3. Physical limitations that impede the patient's ability to participate (e.g., ability to stand),
4. Acute infections or hematuria,
5. Pregnant or actively trying to conceive,
6. History of pelvic irradiation,
7. Concurrent medications with α-adrenergic antagonists or diuretics
8. Pelvic organ prolapse stage III or IV,
9. Severe urethral sphincter weakness and/or defect,
10. Suspected urethral and/or vesical fistula

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Improvement in severity of involuntary urine loss | Baseline, 6 weeks
  Measured by pad testing

SECONDARY OUTCOMES:
incontinence episode frequency | Baseline, 6 weeks
  Daily Diary
health-related quality of life | Baseline, 6 weeks
  Quality of Life questionarie

CONTACTS AND LOCATIONS:
Overall Officials: Nissrine Nakib, MD, Principal Investigator — University of Minnesota
Locations (4):
- United States (4):
  - University of Minnesota Medical Center, Maple Grove, Minnesota
  - Metro OBGYN, Maplewood, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nakib N, Sutherland S, Hallman K, Mianulli M, R Boulware D. Randomized trial of mechanotherapy for the treatment of stress urinary incontinence in women. Ther Adv Urol. 2024 Feb 6;16:17562872241228023. doi: 10.1177/17562872241228023. eCollection 2024 Jan-Dec. PMID 38328552